CLINICAL TRIAL: NCT04272814
Title: Initiating Early Compression Therapy in the Treatment of Lower Limb Cellulitis for Adults Admitted to the Acute Hospital to Improve Patient outcomes-a Feasibility Study
Brief Title: Compression Therapy for Acute Lower Limb Cellulitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The patient pathway changed resulting in less admissions for this condition.
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17/P/203
Record Dates: First submitted 2018-01-15; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Lower Limb Cellulitis

STUDY DESIGN:
Intervention Model Description: compression therapy vs standard therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Compression therapy (Experimental): compression therapy
  Interventions: Other: Compression therapy; Diagnostic Test: initial clinical assessment
- Standard treatment (Active Comparator): standard treatment
  Interventions: Diagnostic Test: initial clinical assessment

INTERVENTIONS:
Other: Compression therapy — Compression application
  Arms: Compression therapy
Diagnostic Test: initial clinical assessment — Initial clinical assessment (includes history, vascular assessment, limb examination and wound assessment where necessary)

SUMMARY:
Initiating early compression therapy in the treatment of lower limb cellulitis for adults admitted to the acute hospital to improve patient outcomes - a pilot study

Cellulitis is a skin infection that results in oedema (additional fluid within tissues), erythema (redness) and variable levels of skin damage. Patients generally present with malaise, pain and if a lower limb is affected they have difficulty mobilising and weight bearing. Patients within this organisation are often referred to the tissue viability service only after significant skin damage has occurred (even thought they are receiving appropriate antibiotic therapy). At this point they will be offered an established plan of care that includes compression therapy if it can be tolerated however at present less than 50% of those being admitted are referred.

Despite compression therapy being well proven in oedema management there is no data available to support or reject the early application in lower limb cellulitis. There is also a lack of information about the impact of early intervention in quality of life for patients in this specific group.

This study has been developed in order to determine the feasibility of being able to undertake a wider trial which would evaluate the outcomes of patients with acute lower limb cellulitis treated with compression therapy versus standard care.

The objectives of the study would be to test the procedures and data collection tools being considered for use in a wider study. This would include collection of quality outcome questionnaires, limb circumference measurements and photography as well as recruitment of participants, the follow up processes and participant attrition. Secondary objectives would be linked to quality of life outcome measures and would determine oedema reduction (and its impact on quality of life), the average number of beddays compared to a historical cohort and to determine recurrence within the study period.

DETAILED DESCRIPTION:
Cellulitis is a skin infection that results in oedema (additional fluid within tissues), erythema (redness) and variable levels of skin damage. Patients generally present with malaise, pain and if a lower limb is affected they have difficulty mobilising and weight bearing. Patients within this organisation are often referred to the tissue viability service only after significant skin damage has occurred (even thought they are receiving appropriate antibiotic therapy). At this point they will be offered an established plan of care that includes compression therapy if it can be tolerated however at present less than 50% of those being admitted are referred.

Despite compression therapy being well proven in oedema management there is no data available to support or reject the early application in lower limb cellulitis. There is also a lack of information about the impact of early intervention in quality of life for patients in this specific group.

This study has been developed in order to determine the feasibility of being able to undertake a wider trial which would evaluate the outcomes of patients with acute lower limb cellulitis treated with compression therapy versus standard care.

The objectives of the study would be to test the procedures and data collection tools being considered for use in a wider study. This would include collection of quality outcome questionnaires, limb circumference measurements and photography as well as recruitment of participants, the follow up processes and participant attrition. Secondary objectives would be linked to quality of life outcome measures and would determine oedema reduction (and its impact on quality of life), the average number of beddays compared to a historical cohort and to determine recurrence within the study period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical features of acute class 2-4 cellulitis of the lower leg
* They have an Ankle Brachial Pressure Index between ≥0.8 and ≤1.3 or Toe Brachial Pressure Index ≥ 0.7 for treatment with full compression therapy
* They have a Laboratory Risk Indicator for Necrotising Fasciitis (LRINEC) score of less than 6 and no clinical signs of necrotising fasciitis
* They are able to tolerate compression therapy, keeping the bandages in place above the level of visible cellulitis for the treatment period
* 18 years or older capable of giving informed consent
* They are admitted to the study setting

Exclusion Criteria:

* Clinical signs or symptoms of peripheral arterial disease
* Unable to give informed consent
* Unable/unwilling to wear compression bandages for study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Recruiting 40 participants within 6 months | 6 months
  Recruitment of 40 participants within 6 months, who meet the eligibility criteria

SECONDARY OUTCOMES:
Determine changes in quality of life outcome measures using EQ-5D-5L questionnaires. | 6 months
  Quality of life outcome measures analysing EQ-5D-5L questionnaires.
Determine oedema reduction. | 6 months
  Measuring limb circumference sequentially to estimate limb volume at each bandage change. Measurement in centimetres.
Determine average number of bed days. | 6 months
  Comparing historical cohort of 40 patients admitted for treatment from April 2017
To determine cellulitis recurrence in patients within the study period. | 6 months
  To record cellulitis recurrence in the 40 patients admitted for treatment from April.

CONTACTS AND LOCATIONS:
Locations (1):
- Derriford Hospital, Plymouth, United Kingdom